CLINICAL TRIAL: NCT05564494
Title: The Arthroscopic Treatment of Anterior Shoulder Instability (ATRASI): A Pilot Multicentre Randomized Controlled Trial
Brief Title: Surgical Treatment of Recurrent Shoulder Dislocations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ivan Wong, MD, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50028
Record Dates: First submitted 2022-09-15; First posted 2022-10-03 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Instability
Keywords: Arthroscopy; Shoulder Instability; Multiple Dislocations

STUDY DESIGN:
Intervention Model Description: This study is a pilot multi-center, double-blinded, RCT of a minimum of 100 patients, performed in five cities at seven sites (Calgary (2 sites), Winnipeg (2 sites), Montreal, Halifax, and Ottawa).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bankart Repair (Active Comparator): Arthroscopic Bankart repair procedures will be performed according to each individual surgeon's usual technique. Procedures will be performed with the patient in the lateral or beach-chair position. Repairs for associated or conjoined superior labral anterior-to-posterior (SLAP) tears will be documented and performed at the surgeon's discretion. Labral detachments will be repaired with the use of suture-anchor fixation and arthroscopic tying techniques. Either two or three suture anchors will be used. Capsular redundancy will be addressed with arthroscopic suture plication at the surgeon's discretion. Surgeons will mobilize the capsulolabral tissue as deemed necessary. Surgical time and video of the operation will be recorded, and photographs will be taken documenting any bone loss.
  Interventions: Procedure: Bankart Repair
- Anatomic Glenoid Reconstruction (Experimental): The surgical technique was the lateral decubitus all-arthroscopic anatomic glenoid reconstruction procedure for treatment of anterior shoulder instability as described by Wong et al. (2015). The procedure is done in a semi-lateral decubitus position that assists with optimal graft placement on the native glenoid. The investigators utilize the cannulated Bristow-Latarjet Instability Shoulder System (Depuy-Mitek, MA, USA). The surgical technique is identical to that of arthroscopic Bankart repair with one additional step. Prior to insertion of anchors, one additional medal portal is created for insertion of the bone graft. The distal tibia allograft is prepared; the cannulated guide is attached and advanced through the rotator interval and secured with two cannulated screws. Finally, the Bankart repair is performed above the graft. Surgical time and video of the operation will be recorded, and photographs will be taken documenting any bone loss.
  Interventions: Procedure: Anatomic Glenoid Reconstruction

INTERVENTIONS:
Procedure: Bankart Repair — Patients Randomized to Bankart Repair Group
  Other Names: Arthroscopic bankart repair
  Arms: Bankart Repair
Procedure: Anatomic Glenoid Reconstruction — Patients Randomized to Anatomic Glenoid Reconstruction Group
  Other Names: Arthroscopic distal tibia bone graft
  Arms: Anatomic Glenoid Reconstruction

SUMMARY:
This is a pilot multi-centre, double blinded randomized controlled trial. The primary outcome of this pilot trial will be feasibility. Prior to conducting a large definitive trial, the investigators will conduct this pilot trial comparing arthroscopic Bankart repair with arthroscopic anatomic glenoid reconstruction (AAGR), evaluating recurrent dislocation rates and functional outcomes over a 24-month period. The feasibility objectives are: (1) to evaluate the investigators ability to recruit patients across multiple sites and (2) to assess study protocol adherence and ability to follow patients to 24 months. Clinical objectives for the pilot trial are exploratory only. The investigators wish to gather means and standard deviations for clinical outcomes to power their future definitive trial. The objectives of the definitive trial will include a comparison of patient-reported outcomes at the two-year post-operative time point, differences in recurrence rates, complication rates, functional shoulder assessments, and return to work/sport.

DETAILED DESCRIPTION:
The glenohumeral joint has the greatest range of motion of any major articulation in the human body. This increased mobility leaves the joint vulnerable to dislocation and the development of instability and osteoarthritis, both of which can have drastic effects on work productivity and quality of life. Symptomatic instability following anterior glenohumeral dislocation is especially common among young people. In patients under 20 years of age, recurrent dislocation rates may be as high as 90%. The high incidence of recurrent dislocation negatively affects the individual and society in general. It may limit range of movement and can require multiple hospital visits for treatment and surgical procedures to prevent further dislocations. Chronic instability of the joint may prevent the individual from participating in sports and physical activity, and from returning to work, and leads to osteoarthritis. The development of osteoarthritis in young patients is devastating and leads to changes within the shoulder that are not easily repairable and results in the need for early shoulder replacements which are costly for both the healthcare system and for the patient themselves. It has been well-established in the literature that surgical management of anterior shoulder instability provides a lower recurrence rate and better rates of return to sport than non-operative treatment. Non-operative treatment of primary anterior shoulder instability has been found to have a high rate of progression to arthritis at a long term follow-up, due to recurrence.

Recurrence rates are influenced by multiple factors including age and gender of the patient, contact sport participation, ligamentous laxity, and the bone loss both on the glenoid and humerus. Of these factors, bone loss is the only modifiable factor. Glenoid defects, present in 22% of patients with acute dislocations, are found in 73% of recurrent dislocations. The management of glenoid bone deficiency in shoulder instability has been a challenge to surgeons for many years. Anteroinferior glenoid bone loss is a significant contributor to recurrent instability through alteration of both the glenohumeral joint contact area and congruency of the articular surfaces. Previous researchers outlined the additive effect of humeral and glenoid bone loss in contributing to shoulder instability and stressed the importance of bony procedures in creating a stable shoulder, particularly for the young active patient. For patients with large anterior glenoid defects (>25%) or other risk factors for recurrence, bone grafting procedures, including autogenous coracoid transfer to the anterior glenoid (i.e. Latarjet procedure) as well as iliac crest autograft and tibial allografts (i.e. arthroscopic anatomic glenoid reconstruction (AAGR)) have been described. These procedures have all been shown to be equally effective and reliable techniques for treating shoulder instability.

The most common pathology in recurrent shoulder instability is anteroinferior capsulolabral avulsion. In 1938, Bankart described the detachment of the anterior inferior labrum from the glenoid rim as a cause of anterior instability and presented his case report of 27 patients treated surgically. In recent years, technical advancements in arthroscopic shoulder surgery have radically altered the treatment of anterior shoulder instability. Arthroscopic techniques have been developed in an attempt to reduce common challenges of open repair including wide dissection, loss of external rotation and post-operative pain. Arthroscopic labral repair, now considered routine and reliable, is the treatment of choice for many cases of recurrent anterior shoulder instability in North America.

Although the results of arthroscopic anterior labral repair using current techniques have been shown to parallel results of open anterior stabilizations in most patients, it is recognized that arthroscopic labral repair is less effective in patients with risk factors for failure such as young age, hyperlaxity, competitive contact sport participation, and in particular glenoid or humeral bone loss. A recently published long-term study on patient outcomes following isolated arthroscopic Bankart repair found a high rate of recurrence and development of arthritis at a 9-12- year follow-up. The authors state that an isolated Bankart repair does not solve the issue of glenoid bone loss.

While bony procedures have traditionally been reserved for cases with bone loss of the glenoid or humerus (so-called Hill-Sachs lesions), there are some regions in which surgeons prefer this type of procedure regardless of the degree of bone loss. This is in part due to recent findings revealing that bone loss may be underestimated by current methods of preoperative measurement. Currently, there are three common methods used to assess bone loss. Preoperative CT and MRI are employed to quantify bone defects, and arthroscopic evaluation may also be used.

There is much controversy over the most accurate method of quantifying bone loss. CT evaluation of glenoid bone loss pre-operatively has been shown to underestimate bone loss.. The absence of a validated non-invasive pre-operative imaging modality has led many surgeons to utilize bony procedures more aggressively, despite limited findings of bone loss on pre-operative imaging. One survey revealed that, irrespective of the types of patients and lesions, 72% of French shoulder surgeons prefer bone block procedures for treating traumatic recurrent anterior shoulder instability. This is in stark contrast to the findings of a large international survey, in which 90% of shoulder surgeons in other countries preferred arthroscopic Bankart repair. Rates of recurrence after these two techniques vary widely in the literature, ranging from 0% to 30% for arthroscopic Bankart repair, with a mean of 9%, and from 2% to 14% for the open Latarjet bone block procedure, with a mean of 7%.

In recent years, trends toward minimally invasive shoulder surgery along with improvements in technology and technique have led surgeons to expand the application of arthroscopic treatment. Techniques have been developed to treat severe instability with or without associated bone loss using arthroscopic bone allograft and autograft augmentation. These approaches seek to provide a nearly anatomic reconstruction of the glenohumeral joint by treating the soft tissue and the bony lesions. Advantages of an arthroscopic approach include smaller incisions, less disruption of the subscapularis, and the ability to evaluate the joint for other intra-articular lesions. The view afforded by the camera may allow for more accurate placement of the graft in the joint.

Rates of instability recurrence after Bankart and bone block procedures vary widely in the literature, ranging from 0% to 30% for arthroscopic Bankart repair and from 2% to 14% for the bone block procedures . A recent systematic review cites the recurrence rates for these two procedures to be 19.5% and 8.7%, respectively. Patients with recurrent dislocations and 25% bone loss make up the majority of instability patients, as opposed to first-time dislocators and patients with >25% bone loss. There is no consensus on the best treatment type for patients with recurrent anterior shoulder instability with subcritical (<25%) bone loss. However, most of the evidence to support bone grafting over soft tissue repair in this patient population has been retrospective, and there has been no randomized controlled trial comparing Bankart with a bone block technique, data regarding newer arthroscopic bony glenoid augmentation is even more limited.

While a multi-site, double-blinded-randomized controlled trial would provide the best evidence for the preferred technique, the feasibility of such a project is unknown. The investigators therefore propose a pilot multi-site, double-blinded randomized controlled trial to compare the outcomes of arthroscopic Bankart repair with those of arthroscopic Bankart repair plus bony glenoid augmentation (i.e. AAGR). The goal of this pilot is to assess the feasibility of recruiting patients across multiple sites while adhering to study protocols before conducting a definitive RCT which requires more resources (financial and otherwise). Additionally, most of the data on the AAGR technique is from a single surgeon and the investigators need to ensure that the results and outcomes are generalizable across multiple surgeons and multiple sites.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent anterior glenohumeral dislocation (two or more incidents)
* Presence of glenoid and/or humerus bone loss on imaging (x Ray, CT or MRI)

Exclusion Criteria:

* Uncontrolled diabetes (Hgb A1C >7%)
* Prior surgery of affected shoulder
* Pregnancy
* Multidirectional instability
* Posterior instability
* Paralysis of the shoulder
* Cancer
* Severe systemic illness
* Presence of massive rotator cuff tear
* Patients that present with < 10% or > 25% bone loss under preoperative imaging.
* Generalized laxity (>5/9 Beighton Score)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Subject Recruitment | Measured throughout the entire study, up to 2 years
  Recruitment of 100 participants
Participant Adherence | Measured throughout the entire study, up to 2 years
  Protocol adherence
Patient Follow-up | Measured throughout the entire study, up to 2 years
  Proportion of Patients Followed at 24 months

SECONDARY OUTCOMES:
The Western Ontario Shoulder Instability Index (WOSI) | Measured at 6 month, 1 year, and 2 year time points
  This questionnaire is used to measure shoulder related quality of life in the participants. The range of possible scores is 0-100, with 0 representing no deficits and 100 representing the worst deficits.
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form | Measured at 6 month, 1 year, and 2 year time points
  This questionnaire is used to evaluate shoulder function, the possible range of scores is 0-100, with 0 representing the best score and 100 representing the worst score.
Disabilities of the Arm, Shoulder, and Hand (DASH) | Measured at 6 month, 1 year, and 2 year time points
  This is a questionnaire used to measure the physical function of the participants, scores range from 0-100 with 0 being the best score and 100 being the worst score possible.
MARX Physical Activity Questionnaire | Measured at 6 month, 1 year, and 2 year time points
  This questionnaire is used to assess the physical activity status of the participants, the possible scores range from 0-16 with 16 being the best possible score.
Quality of Life Assessment (EQ-5D-5L) | Measured at 6 month, 1 year, and 2 year time points
  This questionnaire is used to assess the quality of life of the participants, possible scores range from 0-25 with 0 being the best possible score and 25 being the worst score.
Strength | Measured at 6 month, 1 year, and 2 year time points
  Measurement of shoulder strength using a handheld dynamometer
Incidence of Recurrence | Measured at 6 month, 1 year, and 2 year time points
  How often a subsequent shoulder dislocation occurs, measured with patient report data
Range of Motion | Measured at 6 month, 1 year, and 2 year time points
  Measurement of shoulder range of motion, measured with handheld goniometer
Radiographic Imaging | Measured with at least one CT and one x-ray at any time point prior to surgery and once post surgery up to a year after the surgery. The post surgical time frames for this imaging may differ depending on booking, availability, and wait times
  Measured by observing CT scans and X-Rays

CONTACTS AND LOCATIONS:
Overall Officials: Ivan H Wong, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No